CLINICAL TRIAL: NCT00910130
Title: Insulin Resistance And End Stage Renal Disease: The Role Of Retinol Binding Protein 4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Giovanni Piotti, MD, Unit Of Nephrology, Dialysis And Transplantation, IRCCS Fondazione Policlinico San Matteo, Pavia Italy
Other Study IDs: RBP4
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Insulin Resistance; Diabetes; End Stage Renal Disease
Keywords: Retinol Binding Protein 4; Insulin Resistance; Diabetes; End Stage Renal Disease; Dialysis; Nutrition
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Subcutaneous adipose tissue

GROUPS / COHORTS (2):
- End Stage Renal Disease: Patients suffering from End Stage Renal Disease on Hemodialysis, without Diabetes
- Control: Healthy people, with normal Renal Function and without Diabetes, matched with "ESRD group" for age, gender, BMI

SUMMARY:
The purpose of this study is to determine whether Retinol binding protein 4 has a role in insulin resistance development in patients suffering from end stage renal disease on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis for "End Stage Renal Disease group"
* Normal Renal Function for "Control group"

Exclusion Criteria:

* Diabetes
* Malnutrition
* Malignancy
* Acute Infection
* Chronic Active Infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients or primary care clinic for "End Stage Renal Disease group;" Blood donors or primary care clinic for "Control group"
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Piotti, MD, Principal Investigator — Unit Of Nephrology, Dialysis And Transpantation, IRCCS Fondazione Policlinico San Matteo, Pavia Italy; Teresa Rampino, MD, Study Director — Unit Of Nephrology, Dialysis And Transpantation, IRCCS Fondazione Policlinico San Matteo, Pavia Italy; Antonio Dal Canton, MD, Study Chair — Unit Of Nephrology, Dialysis And Transpantation, IRCCS Fondazione Policlinico San Matteo, Pavia Italy
Locations (1):
- Giovanni Piotti, Pavia, Italy

REFERENCES:
- [Result] Yang Q, Graham TE, Mody N, Preitner F, Peroni OD, Zabolotny JM, Kotani K, Quadro L, Kahn BB. Serum retinol binding protein 4 contributes to insulin resistance in obesity and type 2 diabetes. Nature. 2005 Jul 21;436(7049):356-62. doi: 10.1038/nature03711. PMID 16034410
- [Result] Graham TE, Yang Q, Bluher M, Hammarstedt A, Ciaraldi TP, Henry RR, Wason CJ, Oberbach A, Jansson PA, Smith U, Kahn BB. Retinol-binding protein 4 and insulin resistance in lean, obese, and diabetic subjects. N Engl J Med. 2006 Jun 15;354(24):2552-63. doi: 10.1056/NEJMoa054862. PMID 16775236